CLINICAL TRIAL: NCT01131208
Title: Gene Expression Profiling Using Paraffin-embedded Tissues and the Nuclease Protection Assay in Diffuse Large B-cell Lymphoma (DLBCL) Treated With CHOP or R-CHOP: An ECOG and SWOG Correlative Study of E4494
Brief Title: Biomarkers in Patients With Diffuse Large B-Cell Lymphoma Treated With Combination Chemotherapy With or Without Rituximab
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000671515; ECOG-E4494T2
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Lymphoma
Keywords: contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; recurrent adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Gene Expression Profiling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: gene expression analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer. It may also help doctors predict how well patients will respond to treatment.

PURPOSE: This research study is studying biomarkers in patients with diffuse large B-cell lymphoma treated with combination chemotherapy with or without rituximab.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify genes predictive of clinical outcome (failure-free survival and overall survival) among patients with diffuse large B-cell lymphoma treated with CHOP or R-CHOP induction on ECOG-E4494 using the nuclease protection assay for measuring gene expression in paraffin-embedded tissue.
* To identify genes that change their prognostic profile with the addition of rituximab to CHOP chemotherapy.

OUTLINE: This is a multicenter study.

Unstained formalin-fixed, paraffin-embedded samples are analyzed for gene expression via nuclease protection assay.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of diffuse large B-cell lymphoma
* Treated with CHOP or R-CHOP on ECOG-E4494

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from patients enrolled on E4402 from whom samples were submitted for research
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-04-21 (Actual); Primary Completion 2010-08-21 (Actual); Study Completion 2010-08-21 (Actual)

PRIMARY OUTCOMES:
Identification of genes predictive of clinical outcome | 1 month
Identification of genes that change their prognostic profile with the addition of rituximab to CHOP chemotherapy | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jane N. Winter, MD, Principal Investigator — Robert H. Lurie Cancer Center